CLINICAL TRIAL: NCT03568708
Title: Primary Ovarian Insufficiency: Phenotype and Optimal Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patty Brisben Foundation For Women's Sexual Health (Other)
Responsible Party: Principal Investigator, Halley Wasserman, Assistant Professor, Division of Endocrinology, University of Cincinnati Department of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FP00000706
Record Dates: First submitted 2018-05-11; First posted 2018-06-26 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Primary Ovarian Insufficiency
Keywords: Primary Ovarian Insufficiency; Hormone Replacement Therapy; Estrogen Deficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Ortho Evra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Participants (No Intervention): The control group will reflect a comparison group similar to the POI patient group. As bone density, body composition, and cognitive domains continue to mature throughout the teenage years, this comparison group will provide an important metric of normal growth and development.
- POI Participants (Experimental): This group will be participants who have been recently diagnosed with POI. In an open-label fashion, participants with POI will receive Transdermal Estrogen(beginning at a dose of 25 μg/patch applied weekly), with the dose increased at 3, 6 12, and 18 months (to 37.5, 50, 75, and 100 µg/patch).
  Interventions: Drug: Transdermal Estrogen

INTERVENTIONS:
Drug: Transdermal Estrogen — In an open-label fashion, participants with POI will receive transdermal estradiol (beginning at a dose of 25 µg/patch applied weekly), with the dose increased at 3, 6 12, and 18 months (to 37.5, 50, 75, and 100 µg/patch).
  Other Names: Estradiol-estradiol patch
  Arms: POI Participants

SUMMARY:
This pilot study will observe the progression of newly diagnosed POI patients physical and psychology outcomes after initiating standard of care HRT treatment in comparison to healthy female control participants' physical and psychology health over 24 months.

DETAILED DESCRIPTION:
Background: Primary ovarian insufficiency (POI) is an enigmatic condition that affects ~1/10,000 women by age 20. Sometimes referred to as "early menopause," POI is characterized by estrogen deficiency among other hormonal abnormalities that resemble the menopause. POI is a serious chronic condition with no cure. The clinical presentation or 'phenotype' in adolescents is not well understood. Health consequences may include delayed or arrested puberty, skeletal losses, and the threat to reproductive health. Both the metabolic and emotional sequelae are substantial, and one of the most concerning is compromised bone health. The optimal hormone replacement therapy (HRT) regimen for these young women is debated and practice varies among health providers. Importantly only sparse data exist to guide clinicians to make evidence-based decisions regarding the management of these patients. If initiated early, HRT may prevent estrogen-associated bone loss.

Impact: Better understanding of POI may lead to improved treatments for this underserved population and have significant implications for the treatment of estrogen deficiency in other populations of adolescents and young women, and for all women going though natural menopause later in life. Little is known about the effects of HRT on bone health, body composition, cognition, and health-related quality of life, especially among adolescents. Understanding how this therapy affects these multiple health outcomes will fill knowledge gaps regarding treatment for young patients with POI, with potential implications for adolescents and young women with estrogen deficiency in other clinical settings. We will define the clinical presentation (i.e., phenotype) of adolescent POI. The pilot data collected will be used in a future application to the National Institutes of Health, to fund a larger trial that builds on observations from this initial study. The information gained from this pediatric model may also provide insights on management of the natural menopause that occurs in all women later in life.

Methods: Ten adolescents with idiopathic POI (i.e., from unexplained causes) will be recruited through the Cincinnati Children's Hospital Medical Center (CCHMC) Teen Health Center, Endocrine or Pediatric/Adolescent Gynecology Clinics. Ten healthy controls will be recruited from the Teen Health Center. Participants with POI will receive transdermal estrogen replacement (beginning at 25 µg/patch applied weekly), with the dose increased at subsequent study visits that will occur at 3, 6, 12, 18, and 24 months. All data collection will take place at the CCHMC Schubert Research Clinic. The investigators will measure bone density of the central skeleton and body composition by dual-energy x-ray absorptiometry. To evaluate the peripheral skeleton, bone and muscle measures will be obtained by peripheral quantitative computed tomography. At each visit, the participants will have blood drawn to measure circulating hormone levels that are characteristically altered in adolescents with POI, along with safety assays. Cognitive functioning will be assessed using standardized tools. Participants will complete quality of life assessments, along with nutrition and physical activity surveys. Lastly, all participants will also complete a detailed medical history and health assessment.

Implications/Future Directions: Once the phenotype of adolescent POI is more clearly defined, a logical next question will be to determine whether negative health outcomes can be prevented or modified. Data from the proposed trial will guide the design of future prospective studies that evaluate the effects of traditional treatments (e.g., HRT), including a longer study to monitor HRT therapy, as well as more experimental treatments (e.g., skeletal agents) that may benefit young women with this rare condition. In addition, findings are expected to open avenues of research for adolescents and women with estrogen deficiency in other clinical settings.

ELIGIBILITY:
Inclusion Criteria for POI patients

The participant must:

1. Be willing to give informed consent/assent
2. Have a diagnosis of POI based on 2 elevated serum follicle stimulating hormone (FSH) levels obtained >1 month apart.
3. Be English-speaking

Exclusion Criteria for POI patients

The participant must not:

1. Have other chronic disease known to affect bone health (e.g., cystic fibrosis, celiac disease, etc.)
2. Have an identified secondary cause of ovarian insufficiency
3. Have POI in the setting of Turner syndrome, Fanconi Anemia, galactosemia, or Perrault syndrome (as associated neurological/medical sequelae could confound baseline measures)
4. Have used medications known to affect bone metabolism over previous 3 months (e.g. anticonvulsants, chronic use of glucocorticoids, Depo-Provera, oral contraceptive pills)
5. Be currently pregnant (to be confirmed by pregnancy testing)

Inclusion Criteria for Healthy Adolescent Control Participants

The participant must:

1. Be similar in age and race group to the idiopathic POI group

   1. Control participants age must be within one year of age from the POI participant at the time of enrollment. Age may be within one year older or one year younger
   2. Race of controls participants will be matched based on race of POI patient participants
2. Have a BMI within 20% of the BMI of the case-matched participant
3. If postmenarchal, will be regularly menstruating (cycles between 21-35 days)

   a. if POI participant is <12.5yrs (mean age of menarche) will match with a pre- menarchal control participant
4. Be English-speaking

Exclusion Criteria for Healthy Adolescent Control Participants

The participant must not:

1. Have a chronic disease, known to affect bone metabolism (e.g., cystic fibrosis, celiac disease, sickle cell disease, inflammatory bowel disease etc.)
2. Be receiving medications known to affect bone metabolism over previous three months (e.g. anticonvulsants, chronic use of glucocorticoids, Depo-Provera, oral contraceptive pills, etc.)
3. Have a learning disability or a developmental delay
4. Be currently taking any selective serotonin reuptake inhibitors (SSRIs), antipsychotics or have any documented problems with anxiety or depression.
5. Be currently pregnant (as confirmed by pregnancy testing)

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Gordon, MD,Msc, Principal Investigator — Boston Children's Hospital and Cincinnati Children's Hospital Medical Center; Halley Wasserman, MD, MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon CM, Kanaoka T, Nelson LM. Update on primary ovarian insufficiency in adolescents. Curr Opin Pediatr. 2015 Aug;27(4):511-9. doi: 10.1097/MOP.0000000000000236. PMID 26087426
- [Background] Nelson LM. Clinical practice. Primary ovarian insufficiency. N Engl J Med. 2009 Feb 5;360(6):606-14. doi: 10.1056/NEJMcp0808697. PMID 19196677
- [Background] Committee opinion no. 605: primary ovarian insufficiency in adolescents and young women. Obstet Gynecol. 2014 Jul;124(1):193-197. doi: 10.1097/01.AOG.0000451757.51964.98. PMID 24945456
- [Background] Sadeghi MR. New hopes for the treatment of primary ovarian insufficiency/premature ovarian failure. J Reprod Infertil. 2013 Jan;14(1):1-2. No abstract available. PMID 23926553
- [Background] Gordon CM, Zemel BS, Wren TA, Leonard MB, Bachrach LK, Rauch F, Gilsanz V, Rosen CJ, Winer KK. The Determinants of Peak Bone Mass. J Pediatr. 2017 Jan;180:261-269. doi: 10.1016/j.jpeds.2016.09.056. Epub 2016 Nov 3. No abstract available. PMID 27816219
- [Background] Bakhsh H, Dei M, Bucciantini S, Balzi D, Bruni V. Premature ovarian insufficiency in young girls: repercussions on uterine volume and bone mineral density. Gynecol Endocrinol. 2015 Jan;31(1):65-9. doi: 10.3109/09513590.2014.958987. Epub 2014 Sep 9. PMID 25203144
- [Background] Popat VB, Calis KA, Vanderhoof VH, Cizza G, Reynolds JC, Sebring N, Troendle JF, Nelson LM. Bone mineral density in estrogen-deficient young women. J Clin Endocrinol Metab. 2009 Jul;94(7):2277-83. doi: 10.1210/jc.2008-1878. Epub 2009 Apr 28. PMID 19401379
- [Result] Zemel BS, Kalkwarf HJ, Gilsanz V, Lappe JM, Oberfield S, Shepherd JA, Frederick MM, Huang X, Lu M, Mahboubi S, Hangartner T, Winer KK. Revised reference curves for bone mineral content and areal bone mineral density according to age and sex for black and non-black children: results of the bone mineral density in childhood study. J Clin Endocrinol Metab. 2011 Oct;96(10):3160-9. doi: 10.1210/jc.2011-1111. Epub 2011 Sep 14. PMID 21917867

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Ovarian Insufficiency (POI) Participants: This group will be participants who have been recently diagnosed with Primary ovarian Insufficiency (POI). In an open-label fashion, participants with POI will receive Transdermal Estrogen (beginning at a dose of 25 μg/patch applied weekly), with the dose increased at 3, 6 12, and 18 months (to 37.5, 50, 75, and 100 µg/patch).
Period: Overall Study
Arm/Group | Control Participants | Primary Ovarian Insufficiency (POI) Participants
Started | 9 | 10
Completed | 8 | 8
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: For these analyses, we included all participants who enrolled in the study.
Groups:
- Primary Ovarian Insufficiency (POI) Participants: This group will be participants who have been recently diagnosed with POI. In an open-label fashion, participants with POI will receive Transdermal Estrogen(beginning at a dose of 25 μg/patch applied weekly), with the dose increased at 3, 6 12, and 18 months (to 37.5, 50, 75, and 100 µg/patch).
- Total: Total of all reporting groups
Arm/Group | Control Participants | Primary Ovarian Insufficiency (POI) Participants | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (0.94) | 16.8 (1.25) | 16.8 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 6 | 6 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.90 (4.78) | 26.37 (6.48) | 26.15 (5.79)
Bone Mineral Density Whole Body less head [Mean (Standard Deviation); unit: Z-score] — A bone mineral density (BMD) Z-score is an age, sex and race specific measurement. Normal BMD Z-scores range from -2.0 to 2.0 with 0.0 representing population mean. Higher Z-scores indicate stronger bone density. Z-scores <-2.0 are considered low bone density for age. Height adjustments are made to account for short stature leading to falsely lower BMD Z-scores.
  Z-score | 0.00 (0.96) | -1.93 (0.84) | -1.02 (1.32)
Bone Mineral Density Lumbar Spine [Mean (Standard Deviation); unit: Z-score] — A bone mineral density (BMD) Z-score is an age, sex and race specific measurement. Normal BMD Z-scores range from -2.0 to 2.0 with 0.0 representing population mean. Higher Z-scores indicate stronger bone density. Z-scores <-2.0 are considered low bone density for age. Height adjustments are made to account for short stature leading to falsely lower BMD Z-scores.
  Z-score | 0.80 (0.76) | -1.80 (1.05) | -0.57 (1.61)
Bone Mineral Density Total Hip [Mean (Standard Deviation); unit: Z-score] — A bone mineral density (BMD) Z-score is an age, sex and race specific measurement. Normal BMD Z-scores range from -2.0 to 2.0 with 0.0 representing population mean. Higher Z-scores indicate stronger bone density. Z-scores <-2.0 are considered low bone density for age. Height adjustments are made to account for short stature leading to falsely lower BMD Z-scores.
  Z-score | 0.83 (0.76) | -0.94 (0.68) | -0.10 (1.15)
Bone Mineral Density Femoral Neck [Mean (Standard Deviation); unit: Z-score] — A bone mineral density (BMD) Z-score is an age, sex and race specific measurement. Normal BMD Z-scores range from -2.0 to 2.0 with 0.0 representing population mean. Higher Z-scores indicate stronger bone density. Z-scores <-2.0 are considered low bone density for age. Height adjustments are made to account for short stature leading to falsely lower BMD Z-scores.
  Z-score | 0.91 (0.68) | -1.12 (0.76) | -0.16 (1.26)
Screen for Child Anxiety Related Disorders (SCARED) [Mean (Standard Deviation); unit: units on a scale] — A 41 item self-report tool to assess for anxiety where each question receives a score of either 0, 1 or 2. Range of scores is 0 to 82. A total score of ≥ 25 may indicate the presence of an Anxiety Disorder. A higher score indicates there are more endorsed symptoms of anxiety
  units on a scale | 17.2 (12.2) | 27.0 (14.9) | 22.4 (14.2)
Children's Depression Inventory-II (CDI-2) [Mean (Standard Deviation); unit: units on a scale] — A 28 item self-report test to assess cognitive, affective and behavioral signs of depression in children and adolescents 7 to 17 years old. Scales include Emotional and Functional Problems, along with subscales of Negative mood/Physical symptoms, Negative Self-Esteem, Interpersonal Problems, and Ineffectiveness. The total score is converted into a T-score (mean=50, standard deviation=10) where a result >64 is considered elevated (range <40 to >90). A higher score indicates there are more endorsed symptoms of depression.
  units on a scale | 51.0 (11.4) | 55.3 (10.9) | 53.3 (11.1)
Child and Adolescent Memory Profile (CHaMP) Total Memory Index [Mean (Standard Deviation); unit: units on a scale] — The ChAMP is a norm-referenced test of memory and learning that was designed for use with children, adolescents, and young adults ranging from 5 through 21 years. The ChAMP includes four subtests that measure verbal and visual memory. The tests are administered by a trained professional. The total memory index score is the composite of these four subtests giving an overall estimate of memory with a mean score of 100, standard deviation of15, and range from 50-150.
  units on a scale | 89.5 (9.1) | 93.7 (11.7) | 91.8 (10.6)
Child Health Questionnaire (CHQ-87) Total Score [Mean (Standard Deviation); unit: units on a scale] — The CHQ-87 is an 87-item self-report survey is designed to measure the physical and psychosocial health of adolescents. The total score ranges from 0-100. Higher scores indicate better quality of life. This instrument is reliable and valid for evaluating aspects of health pertinent across age, gender, health condition, and socioeconomic status in adolescents.
  units on a scale | 76.1 (11.6) | 70.1 (12.3) | 72.9 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dual Energy X-ray Absorptiometry (DXA) Measure of Bone Mineral Density (BMD) of the Lumbar Spine
Description: Change in height adjusted areal BMD Z-score of the lumbar spine from baseline to 24 months within groups. BMI Z-score, calcium intake, vitamin D intake and physical activity were included in the analysis. As DXA BMD Z-scores already include race, age, and sex, these variables were not included in the analysis.
  Z-scores ranging between -2.0 and 2.0 are considered normal. A Z-score <-2.0 is considered low. This analysis considers change in Z-score, therefore a high value reflects a greater increase in BMD Z-score.
Time Frame: Change in bone mineral density and body composition from baseline to 24 months
Population: One POI participant had prior oral contraceptive exposure, no matched control, and did not follow up for subsequent visits. For these reasons it was recommended that her data not be included in the analyses.
Measure: Least Squares Mean (Standard Deviation); unit: Z-score
Groups:
- Control Participants: The control group reflects a comparison group similar to the Primary Ovarian Insufficiency (POI) patient group. As bone density, body composition, and cognitive domains continue to mature throughout the teenage years, this comparison group will provide an important metric of normal growth and development.
- POI Participants: This group includes participants diagnosed with POI who completed the transdermal estrogen titration. In an open-label fashion, participants with POI received Transdermal Estrogen (beginning at a dose of 25 μg/patch applied weekly), with the dose increased at 3, 6 12, and 18 months (to 37.5, 50, 75, and 100 µg/patch).
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
Z-score | 0.228 (0.289) | 0.673 (0.289)

2. Secondary Outcome: Change in Dual Energy X-ray Absorptiometry (DXA) Measure of Bone Mineral Density (BMD) at the Whole Body Less Head, Total Hip, and Femoral Neck
Description: To assess changes in bone mineral density DXA height adjusted BMD Z-scores of the whole body less head, total hip and femoral neck were measured. BMI, calcium intake, vitamin D intake and physical activity were included in the analysis. As DXA BMD Z-scores already include race, age, and sex, these variables were not included in the analysis.
  Z-scores ranging between -2.0 and 2.0 are considered normal. A Z-score <-2.0 is considered low. This analysis considers change in Z-score, therefore a high value reflects a greater increase in BMD Z-score.
Time Frame: baseline to 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Z-score
Groups:
- Control Participants: The control group reflects a comparison group similar to the POI patient group. As bone density, body composition, and cognitive domains continue to mature throughout the teenage years, this comparison group will provide an important metric of normal growth and development.
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
Z-score
  Whole Body Less Head | 0.433 (0.199) | 0.815 (0.198)
  Total Hip | 0.231 (0.170) | 0.370 (0.170)
  Femoral Neck | 0.337 (0.195) | 0.556 (0.196)

3. Secondary Outcome: Change in Volumetric Bone Mineral Density (vBMD) at the Distal Radius as Measured by Peripheral Quantitative Computed Tomography (pQCT)
Description: To assess the appendicular (peripheral) skeleton, pQCT (Stratec XCT 2000, Orthometrix, Inc., White Plains, NY) bone measures were obtained of the non-dominant radius at the 3% and 66% sites. Measurements were acquired with a voxel size of 0.4 mm, slice thickness of 2.3 mm, and scan speed of 25 mm/sec, and analyzed with manufacturer software version 6.
Time Frame: Change from baseline to 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: mg/mm^3
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
mg/mm^3
  3% trabecular volumetric BMD | -1.245 (14.484) | -5.415 (14.638)
  66% cortical volumetric BMD | -0.073 (17.728) | 13.945 (18.178)

4. Secondary Outcome: Anthropometrics
Description: The mean BMI in kg/m^2 is presented for each study group at baseline and at the 24 months follow up visit to show that there was no significant difference between groups nor a significant change in BMI over the duration of the study.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 8 | 8
kg/m^2
  BMI at Baseline | 25.9 (4.78) | 27.01 (6.93)
  BMI at 24 months | 27.64 (6.04) | 27.86 (9.62)

5. Secondary Outcome: Change in Lean Mass as Measured by DXA Body Composition
Description: Lean mass was obtained from the whole body DXA scan. Change in baseline to 24 months was assessed.
Time Frame: Change in lean mass from baseline to 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: kg
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
kg | -0.999 (1.754) | 1.577 (1.753)

6. Secondary Outcome: Change in Symptoms of Anxiety as Measured by Screen for Child Anxiety Related Disorders (SCARED)
Description: A 41 item self-report tool to assess for anxiety where each question receives a score of either 0, 1 or 2. Range of scores is 0 to 82. A total score of ≥ 25 may indicate the presence of an Anxiety Disorder. A higher score indicates there are more endorsed symptoms of anxiety.
Time Frame: Change from SCARED score baseline to 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
score on a scale | 8.339 (7.508) | -1.261 (7.454)

7. Secondary Outcome: Change in Symptoms of Depression as Measured by Child Depression Inventory-II (CDI-II)
Description: A brief self-report test that helps assess cognitive, affective and behavioral signs of depression in children and adolescents 7 to 17 years old. Scales include Emotional and Functional Problems, along with subscales of Negative mood/Physical symptoms, Negative Self-Esteem, Interpersonal Problems, and Ineffectiveness. The total score is converted into a T-score (mean=50, standard deviation=10) where a result >64 is considered elevated. A higher score indicates there are more endorsed symptoms of depression.
Time Frame: Change from CDI-II score from baseline to 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: T-score
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
T-score | 1.246 (5.949) | -1.187 (5.793)

8. Secondary Outcome: Change in Memory as Assessed by the Children and Adolescent Memory Profile (CHAMP) Total Memory Index Score
Description: The ChAMP is a norm-referenced test of memory and learning that was designed for use with children, adolescents, and young adults ranging from 5 through 21 years. The ChAMP includes 4 Subtests of visual and verbal memory to generate a total memory index score as a measure of overall memory. The total memory index score ranges from 50-150 with a mean=100 and standard deviation=15. Higher scores indicating better memory. The data presented here is the change in the total memory index score from baseline visit to the 24 month follow up time.
Time Frame: Change from score from baseline to 24 months
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 8 | 8
score on a scale | 17.203 (5.454) | 24.619 (5.379)

9. Secondary Outcome: Change in Quality of Life as Assessed by the Child Health Questionnaire-Child Self-Report Form (CHQ-CF87)
Description: The CHQ-87 is an 87-item self-report survey is designed to measure the physical and psychosocial health of adolescents. The total score ranges from 0-100. Higher scores indicate better quality of life. This instrument is reliable and valid for evaluating aspects of health pertinent across age, gender, health condition, and socioeconomic status in adolescents.
Time Frame: Change from baseline to 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Participants | POI Participants
Number analyzed (Participants) | 9 | 9
score on a scale | 2.710 (6.028) | 5.686 (5.988)

10. Secondary Outcome: Compliance With Transdermal Estrogen Patch
Description: Participants with primary ovarian insufficiency (POI) were prescribed weekly transdermal estrogen (TDE2) patches and asked to log on a patch calendar when they changed the patch. Patch calendars were reviewed for compliance and weeks where at least one patch was applied were considered to be in compliance. Weeks in compliance generated the numerator whereas total weeks of participation in the study constituted the numerator.
Time Frame: Patch Calendars were collected at 6 months, 12 months, 18 months and 24 months. Data presented is through study completion.
Population: As only participants with POI were prescribed TDE2 patches, we only report data on this cohort.
Measure: Mean (Standard Deviation); unit: percentage of weeks with TDE2 use
Groups:
- POI Cases: This group includes participants diagnosed with POI and returned for follow up visits. Weeks of participation in the study were counted from enrollment to date of last study visit.
Arm/Group | POI Cases
Number analyzed (Participants) | 9
percentage of weeks with TDE2 use | 69 (31.4)

11. Secondary Outcome: Study Medications - Serum Estradiol
Description: Mean serum estradiol levels as measured in participants with POI.
Time Frame: Baseline, 12 months, 24 months
Population: The study was originally designed as a 12 month longitudinal trial. Subjects were given the option to continue for 24 months. One case participant declined the extension. As only participants with POI were prescribed transdermal estradiol patches, we only report data on this cohort.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- POI Cases: This group includes participants diagnosed with POI and returned for follow up visits.
Arm/Group | POI Cases
Number analyzed (Participants) | 9
pg/mL
  Estradiol Baseline | 7.49 (2.93)
  Estradiol 12 month | 55.41 (34.75)
  Estradiol 24 month: number analyzed (Participants) | 8
  Estradiol 24 month | 98.63 (93.96)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to completion of the 24 month visit
Groups:
- POI Participants: This group will be participants who have been recently diagnosed with POI. In an open-label fashion, participants with POI will receive Transdermal Estrogen (beginning at a dose of 25 μg/patch applied weekly), with the dose increased at 3, 6 12, and 18 months (to 37.5, 50, 75, and 100 µg/patch).
  For the reporting of adverse events, we included all participants who were enrolled in the study regardless of whether data on our primary or secondary outcomes were analyzed.
Arm/Group | Control Participants | POI Participants
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 4/9 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Participants (N=9) | POI Participants (N=10)
DVT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (DKA) hospitalization (Endocrine disorders) | 0 (0) | 1 (1)
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Participants (N=9) | POI Participants (N=10)
Pain/irritation at patch site (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Foot injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) — No fracture identified
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Breast Lump (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Fibroglandular tissue, normal ultrasound
Vasovagal Syncope (General disorders) | 0 (0) | 1 (1) — During blood draw
Dental extraction (Surgical and medical procedures) | 0 (0) | 1 (1) — Removal of wisdom teeth
Otoralgia (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Motor Tics (Nervous system disorders) | 0 (0) | 1 (1) — Patient with prior diagnosis of simple motor tics reported increased frequency of these events during course of participation in the study.
Folliculitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (DKA) (Endocrine disorders) | 0 (0) | 1 (1) — Patient with known Type 1 Diabetes treated for DKA in emergency room setting. Did not require hospitalization.
Insulin pump site malfunction (Endocrine disorders) | 0 (0) | 1 (1) — Patient with known Type 1 Diabetes seen in local emergency department for insulin pump site malfunction. Resolved with typical care. She was not in DKA.
Weight loss (General disorders) | 0 (0) | 1 (1)
Tympanoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) — Outpatient procedure for cholesteatoma
Viral Illness (Infections and infestations) | 1 (1) | 0 (0)
Metatarsal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mood Changes (Social circumstances) | 0 (0) | 1 (1) — Experienced when not wearing estrogen patch consistently
Headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Motor Vehicle Accident (General disorders) | 1 (1) | 0 (0)
Abdominal Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excessive menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Menstrual bleeding stopped with norethindrone. Additional cycles were shorter in duration and lighter in flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT03568708/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT03568708/ICF_000.pdf